CLINICAL TRIAL: NCT03082261
Title: Multi-center Prospective Study Determining the Sustainability of Pain Relief and Psychosocial and Functional Responses When Utilizing a Multiple Waveform Enabled Neurostimulator
Acronym: TRIUMPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJM-CIP-10145
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain; Intractable Pain
Keywords: Proclaim Elite 5; Proclaim Elite 7; Prodigy; Prodigy MRI; BurstDR Stimulation; Tonic Stimulation; Multiprogram trial stimulator; Invisible trial system
MeSH Terms: conditions — Chronic Pain; Pain, Intractable

STUDY DESIGN:
Intervention Model Description: Post market, international, multicenter, interventional, prospective, single-arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All enrolled subjects (Other): All subjects enrolled into the study with intent to treat with either a Prodigy, Prodigy MRI, or Proclaim Elite Implantable Pulse Generator (IPG).
  Interventions: Device: Prodigy, Prodigy MRI or Proclaim Elite IPG

INTERVENTIONS:
Device: Prodigy, Prodigy MRI or Proclaim Elite IPG — Subjects will be permanently implanted with either a Prodigy, Prodigy MRI or Proclaim Elite IPG

SUMMARY:
The TRIUMPH study is a post-market, international, multicenter, interventional, prospective, single-arm study intended to evaluate the sustainability of pain control and psychosocial and functional responses utilizing a multiple-waveform enabled neurostimulator in subjects with chronic, intractable pain of the trunk and/or limbs.

DETAILED DESCRIPTION:
TRIUMPH study will utilize the multiprogram trial stimulator or invisible trial system with BurstDR for the trial evaluation period and the Prodigy or Proclaim Elite family of neurostimulators with tonic or BurstDR waveform at permanent implant and follow-up for pain control and improvement of psychosocial function. The follow-up visits will be scheduled at 3, 6, 12, 18, and 24 months post permanent implant

ELIGIBILITY:
Inclusion Criteria:

1. Subject has chronic, intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome and intractable low back and leg pain.
2. Subject has a score of 6 or higher on the numeric rating scale (NRS) for average pain specific to the area(s) of chronic pain being treated over the past 24 hours at the baseline visit.
3. Subject is considered by the Investigator as a candidate for implantation of a spinal cord stimulator system according to the system Instructions For Use.
4. Subject is 18 years of age or older at the time of enrollment.
5. Subject is willing to cooperate with the study requirements including compliance with the regimen and completion of all study visits.
6. Subject has signed and received a copy of the Ethics Committee/Institutional Review Board (EC/IRB) approved informed consent.

Exclusion Criteria:

1. Subject currently has a spinal cord stimulation system implanted.
2. Subject has previously failed spinal cord stimulation (SCS) therapy (either trial system evaluation or permanent implant).
3. Subject has a primary diagnosis of Peripheral Vascular Disease (PVD), Angina Pectoris, or Chronic Migraine.
4. Subject has or plans to have a Peripheral Nerve Stimulation system (PNS), Peripheral Nerve field Stimulation system (PNfS), Dorsal Root Ganglion system (DRG), or implantable infusion pump.
5. Subject is currently participating in another clinical investigation with an active treatment arm.
6. Subject unable to read and/or write.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fahey, Study Director — Abbott
Locations (22):
- United States (11):
  - The CORE Institute, Phoenix, Arizona
  - Tory McJunkin MD, Scottsdale, Arizona
  - Pain Institute of Southern Arizona, Tucson, Arizona
  - Chicago Anesthesia Associates, S.C., Chicago, Illinois
  - Pacific Sports & Spine, Eugene, Oregon
  - St. Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Performance Spine and Sports Physicians, P.C., Pottstown, Pennsylvania
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Carolinas Center for Advanced Management of Pain, Greenville, South Carolina
  - Azalea Orthopedics, Tyler, Texas
  - Advanced Pain Management, Greenfield, Wisconsin
- Canada (2):
  - Royal University Hospital, Saskatoon, Saskatchewan
  - CHA L'Enfant Jesus, Québec
- Kuopio University Hospital, Kuopio, Eastern Finland, Finland
- Neurochirurgische Praxis Neuss, Neuss, North Rhine-Westphalia, Germany
- Italy (2):
  - Fondazione I.R.C.C.S. Instituto Neurologico Carlo Besta, Milan, Lombardy
  - Azienda Ospedaliero Univsitaria Pisana, Pisa, Tuscany
- Spain (4):
  - Hospital Virgin de Rocio, Seville, Andalusia
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza, Aragon
  - Hospital Universitario Puerta de Hierro, Majadahonda
  - Hospital Universitari i Politecnic La Fe, Valencia
- Ensemble Hospitalier de la Cote, Hopital de Morges, Morges, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deer TR, Falowski SM, Moore GA, Hutcheson JK, Pena I, Candido K, Cornidez EG, Fraunberg VUZ, Blomme B, Capobianco RA. Passive Recharge Burst Spinal Cord Stimulation Provides Sustainable Improvements in Pain and Psychosocial Function: 2-year Results From the TRIUMPH Study. Spine (Phila Pa 1976). 2022 Apr 1;47(7):548-556. doi: 10.1097/BRS.0000000000004283. PMID 34812195

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 269 subjects were enrolled at 22 investigational sites. The enrollment of the first subject was on 03 March 2017 and the last subject was on 13 February 2018. The last follow-up visit occurred on 26 August 2020.
Period: Overall Study
Arm/Group | All Enrolled Subjects
Started | 269
Completed | 149
Not Completed | 120
Not completed — Death | 4
Not completed — Implant of dorsal root ganglion stimulation (DRG) device | 1
Not completed — Insurance denial | 1
Not completed — Peripheral lead added | 1
Not completed — Withdrawal by Subject | 40
Not completed — Subject did not meet screening inclusion/exclusion criteria | 2
Not completed — Subject implanted with device other than study device | 1
Not completed — Lost to Follow-up | 14
Not completed — Subject moved to a different state | 1
Not completed — Subject non-compliance | 2
Not completed — Subject participation terminated by investigator | 9
Not completed — Subject participation terminated by sponsor | 4
Not completed — System explant | 19
Not completed — Unable to place lead(s) | 2
Not completed — Unsuccessful trial evaluation period | 19

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Subjects: All subjects enrolled into the study with intent to treat with either a Prodigy, Prodigy MRI, or Proclaim Elite IPG.
  Prodigy, Prodigy MRI or Proclaim Elite IPG: Subjects will be permanently implanted with either a Prodigy, Prodigy MRI or Proclaim Elite IPG
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 269
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 166
  Male | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 7
  United States | 210
  Finland | 12
  Italy | 8
  Switzerland | 1
  Germany | 5
  Spain | 26
Duration of Experiencing Chronic Pain [Mean (Standard Deviation); unit: years] | 9.7 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Pain From Baseline to 6 Months Post-permanent Implant, Assessed by the Numeric Rating Scale (NRS)
Description: The pain NRS consists of 1 question that will be asked by interviewing the subjects. Patients will be asked to rate, from 0 (no pain) to 10 (worst imaginable pain), their average pain over the past 24 hours specific to the area(s) of chronic pain being treated. A higher score indicates greater pain intensity.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 181
score on a scale
  Baseline | 7.6 (1.1)
  6 months | 4.6 (2.4)
  Change from baseline to 6 months | 3.0 (2.6)

2. Secondary Outcome: Mean Change in Quality of Life From Baseline to 6 Months Post-permanent Implant, Assessed by the EuroQuol-5 Dimensions (EQ5D) Questionnaire
Description: EQ5D is a standardized instrument for use as a measure of health outcome applicable to a wide range of health conditions and treatments. It provides a simple descriptive profile and a single index value for health status. The EQ5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. A visual analog scale (VAS) for health is also included in the measure as a patient-reported estimate of overall health status. EQ5D Index scores range from - 0.594 (min) to 1 (max). An EQ-5D summary index is derived by applying a formula that attaches values (weights) to each of the levels in each dimension. Higher values represent better outcomes.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 180
score on a scale
  Baseline | 0.44 (0.22)
  6 months | 0.65 (0.21)
  Change from baseline to 6 months | 0.21 (0.22)

3. Secondary Outcome: Mean Change in Pain Catastrophizing From Baseline to 6 Months Post-permanent Implant, Assessed by the Pain Catastrophizing Scale (PCS)
Description: The PCS is a validated scale that measures the magnitude of catastrophizing (negative thoughts and feelings while a patient is experiencing pain). Subjects answer questions about how they feel and what they think about when they are in pain (i.e., not at the current moment). The scale includes 13 statements concerning pain experiences that are rated on a scale between 0 'not at all' and 4 'always'. The scale is self-administered and takes 5 minutes to complete. A higher score indicated a higher level of catastrophizing. PCS total scores range from 0 (min) to 52 (max). Three sub-scales consists of rumination, magnification, and helplessness. Rumination scores range from 0 (min) to 16 (max), Magnification scores range from 0 (min) to 12 (max), and helplessness scores range from 0 (min) to 24 (max). The total PCS score is the sum of the three subscales.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 180
score on a scale
  Baseline | 25.6 (12.9)
  6 months | 13.7 (12.2)
  Change from baseline to 6 months | 11.9 (11.8)

4. Secondary Outcome: Mean Change in Anxiety From Baseline to 6 Months Post-permanent Implant, Assessed by the State-Trait Anxiety Inventory (STAI)
Description: The State-Trait Anxiety inventory is a self-administered screening for anxiety. The STAI has 40 items, 20 items allocated to each of the S-Anxiety and T-Anxiety subscales. All items are rated on a 4-point scale from 1 to 4. It clearly differentiates between the temporary condition of "state anxiety" and the more general and long-standing quality of "trait anxiety" by providing a score for each. Higher scores suggest greater levels of anxiety. The range of possible scores for the STAI varies from a minimum score of 20 to a maximum score of 80 on both the trait and state subscales. The total score is the sum of the two subscales. STAI total scores range from 40 to 160.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 180
score on a scale
  Baseline | 87.1 (26.1)
  6 months | 77.1 (24.7)
  Change from baseline to 6 months | 10.0 (21.6)

5. Secondary Outcome: Mean Change in Depression From Baseline to 6 Months Post-permanent Implant, Assessed by the Patient Health Questionnaire-9 (PHQ9)
Description: The PHQ9 is a multipurpose, validated instrument for screening, diagnosing, monitoring and measuring the severity of depression. The questionnaire consists of 9 questions that rate the frequency of the symptoms of depression. A follow up non-scored question screens and assigns weight to the degree to which depressive problems have affected the patient's level of function. The responses range between 4 choices (0=not at all to 3=nearly every day). Higher scores indicate a higher likelihood of major depression. PHQ-9 scores range from 0 (min) to 27 (max).
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 180
score on a scale
  Baseline | 10.5 (6.5)
  6 months | 7.6 (6.5)
  Change from baseline to 6 months | 3.0 (5.5)

6. Secondary Outcome: Mean Change in Fear Avoidance From Baseline to 6 Months Post-permanent Implant, Assessed by the Tampa Scale for Kinesiophobia (TSK)
Description: The TSK is a 11-item self-report checklist using a 4-point Likert scale that was developed from the original 17-item checklist (Miller, Kopri & Todd, 1991) as a measure of fear or movement or (re)injury. The scale is based on the model of fear avoidance, fear of work related activities, fear of movement and fear of re-injury. The TSK has also been linked to elements of catastrophic thinking. The scale can be useful in measuring unhelpful thoughts and beliefs about pain in people with chronic pain. Total TSK-11 scores range from 11-44 points. Higher scores represent worse outcomes.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 180
score on a scale
  Baseline | 28.7 (7.8)
  6 months | 24.9 (7.2)
  Change from baseline to 6 months | 3.8 (6.7)

7. Secondary Outcome: Mean Change in Sleep From Baseline to 6 Months Post-permanent Implant, Assessed by the Medical Outcome Study (MOS) Sleep Scale
Description: The MOS sleep scale is intended to assess the extent of sleep problems and measures 6 dimensions of sleep, including initiation, maintenance, quantity, adequacy, drowsiness and respiratory impairments. It includes 12 questions with the first question assessing how long it takes the subject to fall asleep. The second question asks how many hours each night the subject slept. The remaining 10 questions have a range of 6 responses from 1="all of the time" to 6="none of the time". The scale is self-administered and validated. MOS Sleep scale scores range from 0 (min) to 100 (max). Higher scores represent worse outcomes.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 180
score on a scale
  Baseline | 52.6 (21.8)
  6 months | 45.0 (23.2)
  Change from baseline to 6 months | 7.5 (18.8)

8. Secondary Outcome: Mean Change in Physical Function From Baseline to 6 Months Post-permanent Implant, Assessed by the Patient-Reported Outcome Measure Information System (PROMIS) Physical Function Scale
Description: The PROMIS Physical Function short form is an 8-item instrument designed to measure physical capability rather than actual performance of physical activities. The scale measures universal physical function rather than disease-specific impairment and assesses current function rather than function over a specified time period. Each question has five potential response options ranging in value from one to five to give a total score ranging from 8 to 40. Scores are converted into t-scores where the average for the general US population is 50 and the SD is 10. Higher scores indicate better physical function.
Time Frame: Baseline to 6 Months
Population: The number of participants analyzed includes subjects who were available at the time of analysis
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 171
T-score
  Baseline | 32.9 (5.0)
  6 months | 36.7 (6.8)
  Change from baseline to 6 months | 3.8 (5.4)

9. Other Pre Specified Outcome: Mean Change in Quality of Life From Baseline to 12 Months Post-permanent Implant, Assessed by the EuroQuol-5 Dimensions (EQ5D) Questionnaire
Description: as for outcome 2
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 162
score on a scale
  Baseline | 0.44 (0.21)
  12 months | 0.63 (0.23)
  Change from baseline to 12 months | 0.20 (0.23)

10. Other Pre Specified Outcome: Mean Change in Quality of Life From Baseline to 18 Months Post-permanent Implant, Assessed by the EuroQuol-5 Dimensions (EQ5D) Questionnaire
Description: as for outcome 2
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 116
score on a scale
  Baseline | 0.44 (0.21)
  18 months | 0.65 (0.20)
  Change from baseline to 18 months | 0.22 (0.23)

11. Other Pre Specified Outcome: Mean Change in Quality of Life From Baseline to 24 Months Post-permanent Implant, Assessed by the EuroQuol-5 Dimensions (EQ5D) Questionnaire
Description: as for outcome 2
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
score on a scale
  Baseline | 0.44 (0.21)
  24 months | 0.64 (0.21)
  Change from baseline to 24 months | 0.21 (0.23)

12. Other Pre Specified Outcome: Mean Change in Pain Catastrophizing From Baseline to 3 Months Post-permanent Implant, Assessed by the Pain Catastrophizing Scale (PCS)
Description: as for outcome 3
Time Frame: Baseline to 3 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 192
score on a scale
  Baseline | 25.7 (13.1)
  3 months | 14.6 (12.3)
  Change from baseline to 3 months | 10.6 (13.4)

13. Other Pre Specified Outcome: Mean Change in Pain Catastrophizing From Baseline to 12 Months Post-permanent Implant, Assessed by the Pain Catastrophizing Scale (PCS)
Description: as for outcome 3
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 162
score on a scale
  Baseline | 25.7 (13.1)
  12 months | 14.3 (13.1)
  Change from baseline to 12 months | 11.3 (12.1)

14. Other Pre Specified Outcome: Mean Change in Pain Catastrophizing From Baseline to 18 Months Post-permanent Implant, Assessed by the Pain Catastrophizing Scale (PCS)
Description: as for outcome 3
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 116
score on a scale
  Baseline | 25.7 (13.1)
  18 months | 14.0 (11.5)
  Change from baseline to 18 months | 12.4 (12.8)

15. Other Pre Specified Outcome: Mean Change in Pain Catastrophizing From Baseline to 24 Months Post-permanent Implant, Assessed by the Pain Catastrophizing Scale (PCS)
Description: as for outcome 3
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
score on a scale
  Baseline | 25.7 (13.1)
  24 months | 13.2 (12.6)
  Change from baseline to 24 months | 12.5 (12.8)

16. Other Pre Specified Outcome: Mean Change in Anxiety From Baseline to 12 Months Post-permanent Implant, Assessed by the State-Trait Anxiety Inventory (STAI)
Description: as for outcome 4
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 162
score on a scale
  Baseline | 87.5 (26.2)
  12 months | 77.3 (26.9)
  Change from baseline to 12 months | 9.3 (22.2)

17. Other Pre Specified Outcome: Mean Change in Anxiety From Baseline to 18 Months Post-permanent Implant, Assessed by the State-Trait Anxiety Inventory (STAI)
Description: as for outcome 4
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 116
score on a scale
  Baseline | 87.5 (26.2)
  18 months | 75.1 (24.9)
  Change from baseline to 18 months | 11.4 (21.4)

18. Other Pre Specified Outcome: Mean Change in Anxiety From Baseline to 24 Months Post-permanent Implant, Assessed by the State-Trait Anxiety Inventory (STAI)
Description: as for outcome 4
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
score on a scale
  Baseline | 87.5 (26.2)
  24 months | 75.5 (26.7)
  Change from baseline to 24 months | 10.8 (21.7)

19. Other Pre Specified Outcome: Mean Change in Depression From Baseline to 12 Months Post-permanent Implant, Assessed by the Patient Health Questionnaire-9 (PHQ9)
Description: as for outcome 5
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 162
score on a scale
  Baseline | 10.2 (6.5)
  12 months | 7.7 (6.6)
  Change from baseline to 12 months | 2.8 (5.6)

20. Other Pre Specified Outcome: Mean Change in Depression From Baseline to 18 Months Post-permanent Implant, Assessed by the Patient Health Questionnaire-9 (PHQ9)
Description: as for outcome 5
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 116
score on a scale
  Baseline | 10.2 (6.5)
  18 months | 6.9 (5.8)
  Change from baseline to 18 months | 3.7 (6.4)

21. Other Pre Specified Outcome: Mean Change in Depression From Baseline to 24 Months Post-permanent Implant, Assessed by the Patient Health Questionnaire-9 (PHQ9)
Description: as for outcome 5
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
score on a scale
  Baseline | 10.2 (6.5)
  24 months | 7.5 (6.4)
  Change from baseline to 24 months | 3.0 (6.1)

22. Other Pre Specified Outcome: Mean Change in Fear Avoidance From Baseline to 3 Months Post-permanent Implant, Assessed by the Tampa Scale for Kinesiophobia (TSK)
Description: as for outcome 6
Time Frame: Baseline to 3 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 191
score on a scale
  Baseline | 28.7 (7.7)
  3 months | 24.6 (7.2)
  Change from baseline to 3 months | 3.8 (7.5)

23. Other Pre Specified Outcome: Mean Change in Fear Avoidance From Baseline to 12 Months Post-permanent Implant, Assessed by the Tampa Scale for Kinesiophobia (TSK)
Description: as for outcome 6
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 162
score on a scale
  Baseline | 28.7 (7.7)
  12 months | 24.4 (7.2)
  Change from baseline to 12 months | 4.3 (7.1)

24. Other Pre Specified Outcome: Mean Change in Fear Avoidance From Baseline to 18 Months Post-permanent Implant, Assessed by the Tampa Scale for Kinesiophobia (TSK)
Description: as for outcome 6
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 116
score on a scale
  Baseline | 28.7 (7.7)
  18 months | 24.3 (7.4)
  Change from baseline to 18 months | 4.8 (7.5)

25. Other Pre Specified Outcome: Mean Change in Fear Avoidance From Baseline to 24 Months Post-permanent Implant, Assessed by the Tampa Scale for Kinesiophobia (TSK)
Description: as for outcome 6
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 139
score on a scale
  Baseline | 28.7 (7.7)
  24 months | 25.2 (7.5)
  Change from baseline to 24 months | 4.2 (7.6)

26. Other Pre Specified Outcome: Mean Change in Sleep From Baseline to 12 Months Post-permanent Implant, Assessed by the Medical Outcome Study (MOS) Sleep Scale
Description: as for outcome 7
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 162
score on a scale
  Baseline | 50.3 (22.6)
  12 months | 45.4 (23.5)
  Change from baseline to 12 months | 7.6 (20.0)

27. Other Pre Specified Outcome: Mean Change in Sleep From Baseline to 18 Months Post-permanent Implant, Assessed by the Medical Outcome Study (MOS) Sleep Scale
Description: as for outcome 7
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 116
score on a scale
  Baseline | 50.3 (22.6)
  18 months | 43.8 (23.8)
  Change from baseline to 18 months | 9.9 (20.6)

28. Other Pre Specified Outcome: Mean Change in Sleep From Baseline to 24 Months Post-permanent Implant, Assessed by the Medical Outcome Study (MOS) Sleep Scale
Description: as for outcome 7
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 139
score on a scale
  Baseline | 50.3 (22.6)
  24 months | 43.2 (22.1)
  Change from baseline to 24 months | 10.8 (20.7)

29. Other Pre Specified Outcome: Mean Change in Physical Function From Baseline to 12 Months Post-permanent Implant, Assessed by the Patient-Reported Outcome Measure Information System (PROMIS) Physical Function Scale
Description: as for outcome 8
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 155
T-score
  Baseline | 33.0 (5.2)
  12 months | 36.3 (6.6)
  Change from baseline to 12 months | 3.2 (5.4)

30. Other Pre Specified Outcome: Mean Change in Physical Function From Baseline to 18 Months Post-permanent Implant, Assessed by the Patient-Reported Outcome Measure Information System (PROMIS) Physical Function Scale
Description: as for outcome 8
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 110
T-score
  Baseline | 33.0 (5.2)
  18 months | 37.1 (6.3)
  Change from baseline to 18 months | 3.7 (6.1)

31. Other Pre Specified Outcome: Mean Change in Physical Function From Baseline to 24 Months Post-permanent Implant, Assessed by the Patient-Reported Outcome Measure Information System (PROMIS) Physical Function Scale
Description: as for outcome 8
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 134
T-score
  Baseline | 33.0 (5.2)
  24 months | 36.9 (7.6)
  Change from baseline to 24 months | 3.8 (6.8)

32. Other Pre Specified Outcome: Mean Change in Pain From Baseline to End of Trial System (Post-permanent Implant), Assessed by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Baseline to end of trial system evaluation, approximately 5 to 7 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 244
score on a scale
  Baseline | 7.7 (1.2)
  End of trial | 3.5 (2.1)
  Change from baseline to end of trial | 4.2 (2.3)

33. Other Pre Specified Outcome: Mean Change in Pain From Baseline to 3 Months Post-permanent Implant, Assessed by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Baseline to 3 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 192
score on a scale
  Baseline | 7.7 (1.2)
  3 months | 4.4 (2.4)
  Change from baseline to 3 months | 3.3 (2.5)

34. Other Pre Specified Outcome: Mean Change in Pain From Baseline to 12 Months Post-permanent Implant, Assessed by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Baseline to 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 163
score on a scale
  Baseline | 7.7 (1.2)
  12 months | 4.7 (2.5)
  Change from baseline to 12 months | 2.9 (2.5)

35. Other Pre Specified Outcome: Mean Change in Pain From Baseline to 18 Months Post-permanent Implant, Assessed by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Baseline to 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 145
score on a scale
  Baseline | 7.7 (1.2)
  18 months | 4.5 (2.5)
  Change from baseline to 18 months | 3.1 (2.6)

36. Other Pre Specified Outcome: Mean Change in Pain From Baseline to 24 Months Post-permanent Implant, Assessed by the Numeric Rating Scale (NRS)
Description: as for outcome 1
Time Frame: Baseline to 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
score on a scale
  Baseline | 7.7 (1.2)
  24 months | 4.8 (2.5)
  Change from baseline to 24 months | 2.8 (2.6)

37. Other Pre Specified Outcome: Number of Participants With Patient Satisfaction at End of Trial System Evaluation
Description: Patient satisfaction will be summarized by count and percentage of participants
Time Frame: End of trial system evaluation, approximately 5 to 7 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 244
Participants
  Very Satisfied | 125
  Satisfied | 94
  Neither Satisfied or Dissatisfied | 7
  Dissatisfied | 10
  Very Dissatisfied | 8

38. Other Pre Specified Outcome: Number of Participants With Patient Satisfaction at 3 Months
Description: Patient satisfaction will be summarized by count and percentage of participants
Time Frame: 3 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 192
Participants
  Very Satisfied | 72
  Satisfied | 75
  Neither Satisfied or Dissatisfied | 31
  Dissatisfied | 14
  Very Dissatisfied | 0

39. Other Pre Specified Outcome: Number of Participants With Patient Satisfaction at 6 Months
Description: Patient satisfaction will be summarized by count and percentage of participants
Time Frame: 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 181
Participants
  Very Satisfied | 67
  Satisfied | 68
  Neither Satisfied or Dissatisfied | 34
  Dissatisfied | 11
  Very Dissatisfied | 1

40. Other Pre Specified Outcome: Number of Participants With Patient Satisfaction at 12 Months
Description: Patient satisfaction will be summarized by count and percentage of participants
Time Frame: 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 163
Participants
  Very Satisfied | 58
  Satisfied | 75
  Neither Satisfied or Dissatisfied | 21
  Dissatisfied | 7
  Very Dissatisfied | 2

41. Other Pre Specified Outcome: Number of Participants With Patient Satisfaction at 18 Months
Description: Patient satisfaction will be summarized by count and percentage of participants
Time Frame: 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 145
Participants
  Very Satisfied | 63
  Satisfied | 57
  Neither Satisfied or Dissatisfied | 17
  Dissatisfied | 7
  Very Dissatisfied | 1

42. Other Pre Specified Outcome: Number of Participants With Patient Satisfaction at 24 Months
Description: Patient satisfaction will be summarized by count and percentage of participants
Time Frame: 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
Participants
  Very Satisfied | 55
  Satisfied | 63
  Neither Satisfied or Dissatisfied | 18
  Dissatisfied | 4
  Very Dissatisfied | 0

43. Other Pre Specified Outcome: Rate of Global Improvement of the Patient by Using the Patient Global Impression of Change (PGIC) at the End of Trial System Evaluation
Description: The PGIC is a categorical rating scale used to evaluate the subject's impression of change in his/her condition since the beginning of the study treatment. The subject rates their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale via an interview technique. The categories are as follows: 1-no change, 2-almost the same, 3-a little better, 4-somewhat better, 5-moderately better, 6-better, and 7-a great deal better. Although this tool does not specify the area of change (e.g., pain, function, quality of life, etc.), it allows for an overall integrated assessment from the prospective of the subject. PGIC values of 6 or 7 are reported to correlate best with actual change.
Time Frame: End of trial system evaluation, approximately 5 to 7 days of BurstDR stimulation
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 244
Participants
  No Change | 18
  Almost the Same | 7
  A little Better | 6
  Somewhat Better | 12
  Moderately Better | 53
  Better | 103
  A Great Deal Better | 45

44. Other Pre Specified Outcome: Rate of Global Improvement of the Patient by Using the Patient Global Impression of Change (PGIC) at 3 Months
Description: as for outcome 43
Time Frame: 3 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 192
Participants
  No Change | 13
  Almost the Same | 12
  A little Better | 20
  Somewhat Better | 22
  Moderately Better | 45
  Better | 50
  A Great Deal Better | 30

45. Other Pre Specified Outcome: Rate of Global Improvement of the Patient by Using the Patient Global Impression of Change (PGIC) at 6 Months
Description: as for outcome 43
Time Frame: 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 181
Participants
  No Change | 12
  Almost the Same | 16
  A little Better | 15
  Somewhat Better | 21
  Moderately Better | 39
  Better | 56
  A Great Deal Better | 22

46. Other Pre Specified Outcome: Rate of Global Improvement of the Patient by Using the Patient Global Impression of Change (PGIC) at 12 Months
Description: as for outcome 43
Time Frame: 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 163
Participants
  No Change | 9
  Almost the Same | 8
  A little Better | 15
  Somewhat Better | 22
  Moderately Better | 34
  Better | 48
  A Great Deal Better | 27

47. Other Pre Specified Outcome: Rate of Global Improvement of the Patient by Using the Patient Global Impression of Change (PGIC) at 18 Months
Description: as for outcome 43
Time Frame: 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 145
Participants
  No Change | 7
  Almost the Same | 10
  A little Better | 11
  Somewhat Better | 8
  Moderately Better | 37
  Better | 47
  A Great Deal Better | 25

48. Other Pre Specified Outcome: Rate of Global Improvement of the Patient by Using the Patient Global Impression of Change (PGIC) at 24 Months
Description: as for outcome 43
Time Frame: 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
Participants
  No Change | 5
  Almost the Same | 4
  A little Better | 12
  Somewhat Better | 13
  Moderately Better | 39
  Better | 40
  A Great Deal Better | 27

49. Other Pre Specified Outcome: Rate of Medication Usage Measured as Number of Participants With Decrease in Chronic Pain Related Medication Intake Since Baseline
Description: Medication usage measured as decrease in chronic pain related medication intake since baseline
Time Frame: 3 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 192
Participants
  Analgesic: number analyzed (Participants) | 113
  Analgesic | 37
  Anti-convulsant: number analyzed (Participants) | 83
  Anti-convulsant | 25
  Muscle Relaxant: number analyzed (Participants) | 33
  Muscle Relaxant | 7
  Non-steroidal Anti-inflammatory Drug: number analyzed (Participants) | 33
  Non-steroidal Anti-inflammatory Drug | 10
  Opioid Medication: number analyzed (Participants) | 154
  Opioid Medication | 60
  Psychiatric Medication: number analyzed (Participants) | 41
  Psychiatric Medication | 10

50. Other Pre Specified Outcome: Rate of Medication Usage Measured as Number of Participants With Decrease in Chronic Pain Related Medication Intake Since Baseline
Description: Medication usage measured as decrease in chronic pain related medication intake since baseline
Time Frame: 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 181
Participants
  Analgesic: number analyzed (Participants) | 110
  Analgesic | 44
  Anti-convulsant: number analyzed (Participants) | 81
  Anti-convulsant | 31
  Muscle Relaxant: number analyzed (Participants) | 31
  Muscle Relaxant | 4
  Non-steroidal Anti-inflammatory Drug: number analyzed (Participants) | 32
  Non-steroidal Anti-inflammatory Drug | 12
  Opioid Medication: number analyzed (Participants) | 147
  Opioid Medication | 62
  Psychiatric Medication: number analyzed (Participants) | 40
  Psychiatric Medication | 11

51. Other Pre Specified Outcome: Rate of Medication Usage Measured as Number of Participants With Decrease in Chronic Pain Related Medication Intake Since Baseline
Description: Medication usage measured as decrease in chronic pain related medication intake since baseline
Time Frame: 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 163
Participants
  Analgesic: number analyzed (Participants) | 102
  Analgesic | 45
  Anti-convulsant: number analyzed (Participants) | 74
  Anti-convulsant | 31
  Muscle Relaxant: number analyzed (Participants) | 31
  Muscle Relaxant | 6
  Non-steroidal Anti-inflammatory Drug: number analyzed (Participants) | 33
  Non-steroidal Anti-inflammatory Drug | 13
  Opioid Medication: number analyzed (Participants) | 128
  Opioid Medication | 61
  Psychiatric Medication: number analyzed (Participants) | 36
  Psychiatric Medication | 11

52. Other Pre Specified Outcome: Rate of Medication Usage Measured as Number of Participants With Decrease in Chronic Pain Related Medication Intake Since Baseline
Description: Medication usage measured as decrease in chronic pain related medication intake since baseline
Time Frame: 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 145
Participants
  Analgesic: number analyzed (Participants) | 95
  Analgesic | 44
  Anti-convulsant: number analyzed (Participants) | 69
  Anti-convulsant | 31
  Muscle Relaxant: number analyzed (Participants) | 26
  Muscle Relaxant | 11
  Non-steroidal Anti-inflammatory Drug: number analyzed (Participants) | 29
  Non-steroidal Anti-inflammatory Drug | 15
  Opioid Medication: number analyzed (Participants) | 115
  Opioid Medication | 60
  Psychiatric Medication: number analyzed (Participants) | 33
  Psychiatric Medication | 16

53. Other Pre Specified Outcome: Rate of Medication Usage Measured as Number of Participants With Decrease in Chronic Pain Related Medication Intake Since Baseline
Description: Medication usage measured as decrease in chronic pain related medication intake since baseline
Time Frame: 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 140
Participants
  Analgesic: number analyzed (Participants) | 89
  Analgesic | 42
  Anti-convulsant: number analyzed (Participants) | 62
  Anti-convulsant | 29
  Muscle Relaxant: number analyzed (Participants) | 24
  Muscle Relaxant | 9
  Non-steroidal Anti-inflammatory Drug: number analyzed (Participants) | 30
  Non-steroidal Anti-inflammatory Drug | 15
  Opioid Medication: number analyzed (Participants) | 108
  Opioid Medication | 51
  Psychiatric Medication: number analyzed (Participants) | 31
  Psychiatric Medication | 14

54. Other Pre Specified Outcome: Number of Participants With Stimulation Sensation Assessed by Stimulation Assessment Form
Description: The Stimulation Assessment Form includes questions to identify the sensations experienced when stimulation is used.
Time Frame: 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 192
Participants
  Burning: number analyzed (Participants) | 108
  Burning | 6
  Buzzing/vibrating/Pulsing: number analyzed (Participants) | 108
  Buzzing/vibrating/Pulsing | 23
  Cold: number analyzed (Participants) | 108
  Cold | 2
  Heaviness: number analyzed (Participants) | 108
  Heaviness | 2
  Itching: number analyzed (Participants) | 108
  Itching | 5
  Massaging/pressure: number analyzed (Participants) | 108
  Massaging/pressure | 3
  Numbness: number analyzed (Participants) | 108
  Numbness | 6
  Stinging/prickling: number analyzed (Participants) | 108
  Stinging/prickling | 6
  Tickling: number analyzed (Participants) | 108
  Tickling | 8
  Tingling: number analyzed (Participants) | 108
  Tingling | 27
  Warm: number analyzed (Participants) | 107
  Warm | 3
  Other: number analyzed (Participants) | 100
  Other | 0

55. Other Pre Specified Outcome: Number of Participants With Stimulation Sensation Assessed by Stimulation Assessment Form
Description: The Stimulation Assessment Form includes questions to identify the sensations experienced when stimulation is used.
Time Frame: 6 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 181
Participants
  Burning: number analyzed (Participants) | 97
  Burning | 3
  Buzzing/vibrating/Pulsing: number analyzed (Participants) | 97
  Buzzing/vibrating/Pulsing | 18
  Cold: number analyzed (Participants) | 97
  Cold | 2
  Heaviness: number analyzed (Participants) | 97
  Heaviness | 4
  Itching: number analyzed (Participants) | 97
  Itching | 2
  Massaging/pressure: number analyzed (Participants) | 97
  Massaging/pressure | 6
  Numbness: number analyzed (Participants) | 97
  Numbness | 9
  Stinging/prickling: number analyzed (Participants) | 97
  Stinging/prickling | 9
  Tickling: number analyzed (Participants) | 97
  Tickling | 6
  Tingling: number analyzed (Participants) | 97
  Tingling | 28
  Warm: number analyzed (Participants) | 97
  Warm | 2
  Other: number analyzed (Participants) | 94
  Other | 0

56. Other Pre Specified Outcome: Number of Participants With Stimulation Sensation Assessed by Stimulation Assessment Form
Description: The Stimulation Assessment Form includes questions to identify the sensations experienced when stimulation is used.
Time Frame: 12 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 163
Participants
  Burning: number analyzed (Participants) | 81
  Burning | 1
  Buzzing/vibrating/Pulsing: number analyzed (Participants) | 81
  Buzzing/vibrating/Pulsing | 13
  Cold: number analyzed (Participants) | 81
  Cold | 1
  Heaviness: number analyzed (Participants) | 80
  Heaviness | 3
  Itching: number analyzed (Participants) | 81
  Itching | 1
  Massaging/pressure: number analyzed (Participants) | 81
  Massaging/pressure | 2
  Numbness: number analyzed (Participants) | 80
  Numbness | 0
  Stinging/prickling: number analyzed (Participants) | 81
  Stinging/prickling | 0
  Tickling: number analyzed (Participants) | 81
  Tickling | 2
  Tingling: number analyzed (Participants) | 81
  Tingling | 19
  Warm: number analyzed (Participants) | 81
  Warm | 1
  Other: number analyzed (Participants) | 79
  Other | 2

57. Other Pre Specified Outcome: Number of Participants With Stimulation Sensation Assessed by Stimulation Assessment Form
Description: The Stimulation Assessment Form includes questions to identify the sensations experienced when stimulation is used.
Time Frame: 18 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 146
Participants
  Burning: number analyzed (Participants) | 73
  Burning | 2
  Buzzing/vibrating/Pulsing: number analyzed (Participants) | 73
  Buzzing/vibrating/Pulsing | 13
  Cold: number analyzed (Participants) | 73
  Cold | 2
  Heaviness: number analyzed (Participants) | 73
  Heaviness | 0
  Itching: number analyzed (Participants) | 73
  Itching | 1
  Massaging/pressure: number analyzed (Participants) | 73
  Massaging/pressure | 4
  Numbness: number analyzed (Participants) | 73
  Numbness | 2
  Stinging/prickling: number analyzed (Participants) | 73
  Stinging/prickling | 2
  Tickling: number analyzed (Participants) | 73
  Tickling | 6
  Tingling: number analyzed (Participants) | 73
  Tingling | 14
  Warm: number analyzed (Participants) | 73
  Warm | 3
  Other: number analyzed (Participants) | 67
  Other | 3

58. Other Pre Specified Outcome: Number of Participants With Stimulation Sensation Assessed by Stimulation Assessment Form
Description: The Stimulation Assessment Form includes questions to identify the sensations experienced when stimulation is used.
Time Frame: 24 Months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 141
Participants
  Burning: number analyzed (Participants) | 55
  Burning | 2
  Buzzing/vibrating/Pulsing: number analyzed (Participants) | 55
  Buzzing/vibrating/Pulsing | 16
  Cold: number analyzed (Participants) | 55
  Cold | 1
  Heaviness: number analyzed (Participants) | 55
  Heaviness | 0
  Itching: number analyzed (Participants) | 55
  Itching | 2
  Massaging/pressure: number analyzed (Participants) | 55
  Massaging/pressure | 7
  Numbness: number analyzed (Participants) | 55
  Numbness | 3
  Stinging/prickling: number analyzed (Participants) | 55
  Stinging/prickling | 3
  Tickling: number analyzed (Participants) | 55
  Tickling | 5
  Tingling: number analyzed (Participants) | 55
  Tingling | 20
  Warm: number analyzed (Participants) | 55
  Warm | 0
  Other: number analyzed (Participants) | 53
  Other | 0

59. Other Pre Specified Outcome: Number of Patient Waveform Preference
Description: Participants could choose between two waveforms with different amplitude, pulse width and frequency to stimulate the spinal cord (burst or tonic). Patient waveform preference post-permanent implant is summarized by counts and percentages.
Time Frame: 3 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 192
Participants
  Burst | 169
  Tonic | 23

60. Other Pre Specified Outcome: Number of Patient Waveform Preference
Description: as for outcome 59
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 181
Participants
  Burst | 158
  Tonic | 23

61. Other Pre Specified Outcome: Number of Patient Waveform Preference
Description: as for outcome 59
Time Frame: 12 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 163
Participants
  Burst | 142
  Tonic | 21

62. Other Pre Specified Outcome: Number of Patient Waveform Preference
Description: as for outcome 59
Time Frame: 18 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 144
Participants
  Burst | 123
  Tonic | 21

63. Other Pre Specified Outcome: Number of Patient Waveform Preference
Description: as for outcome 59
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 139
Participants
  Burst | 116
  Tonic | 23

64. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Frequency of Recharge
Description: Recharging activities throughout the follow-up period for subjects who were implanted with a rechargeable device will be summarized by count and percentage of participants.
Time Frame: 3 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 45
Participants
  2-3 times a week | 8
  Weekly | 24
  Every other week | 6
  Every three week | 3
  Once a month or less often | 4

65. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Frequency of Recharge
Description: as for outcome 64
Time Frame: 6 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 39
Participants
  2-3 times a week | 8
  Weekly | 16
  Every other week | 8
  Every three week | 2
  Once a month or less often | 5

66. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Frequency of Recharge
Description: as for outcome 64
Time Frame: 12 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 32
Participants
  2-3 times a week | 4
  Weekly | 15
  Every other week | 7
  Every three week | 4
  Once a month or less often | 2

67. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Frequency of Recharge
Description: as for outcome 64
Time Frame: 18 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 24
Participants
  2-3 times a week | 3
  Weekly | 13
  Every other week | 5
  Every three week | 1
  Once a month or less often | 2

68. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Frequency of Recharge
Description: as for outcome 64
Time Frame: 24 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 25
Participants
  2-3 times a week | 3
  Weekly | 11
  Every other week | 6
  Every three week | 1
  Once a month or less often | 4

69. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Duration of Recharge
Description: as for outcome 64
Time Frame: 3 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 45
Participants
  Less than 30 Min | 2
  30 Min to 1 Hour | 13
  1 to 2 Hours | 16
  2 to 3 Hours | 9
  3 to 4 Hours | 3
  4 to 5 Hours | 1
  More than 5 Hours | 1

70. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Duration of Recharge
Description: as for outcome 64
Time Frame: 6 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 39
Participants
  Less than 30 Min | 1
  30 Min to 1 Hour | 6
  1 to 2 Hours | 18
  2 to 3 Hours | 7
  3 to 4 Hours | 5
  4 to 5 Hours | 1
  More than 5 Hours | 1

71. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Duration of Recharge
Description: as for outcome 64
Time Frame: 12 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 32
Participants
  Less than 30 Min | 0
  30 Min to 1 Hour | 1
  1 to 2 Hours | 18
  2 to 3 Hours | 7
  3 to 4 Hours | 4
  4 to 5 Hours | 2
  More than 5 Hours | 0

72. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Duration of Recharge
Description: as for outcome 64
Time Frame: 18 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 24
Participants
  Less than 30 Min | 0
  30 Min to 1 Hour | 3
  1 to 2 Hours | 10
  2 to 3 Hours | 7
  3 to 4 Hours | 3
  4 to 5 Hours | 1
  More than 5 Hours | 0

73. Other Pre Specified Outcome: Recharging Activities- Number of Participants With Duration of Recharge
Description: as for outcome 64
Time Frame: 24 months
Population: The number of participants analyzed includes subjects with a rechargeable device
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Subjects
Number analyzed (Participants) | 25
Participants
  Less than 30 Min | 0
  30 Min to 1 Hour | 4
  1 to 2 Hours | 4
  2 to 3 Hours | 9
  3 to 4 Hours | 4
  4 to 5 Hours | 2
  More than 5 Hours | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | All Enrolled Subjects
All-Cause Mortality (participants affected / at risk) | 4/269
Serious Adverse Events (participants affected / at risk) | 18/269
Other Adverse Events (participants affected / at risk) | 27/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=269)
Acute Respiratory Failure with Flash Pulmonary Edema (Injury, poisoning and procedural complications) | 1 (1)
Allergic or Rejection Response to Implant Materials (Injury, poisoning and procedural complications) | 1 (1)
Changes in Stimulation or Reduced Pain Relief Due to Lead Migration (Injury, poisoning and procedural complications) | 2 (2)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Infection (Injury, poisoning and procedural complications) | 5 (5)
Keloid Infection (Injury, poisoning and procedural complications) | 1 (2)
Lead Fracture (Injury, poisoning and procedural complications) | 1 (1)
Oversedation (Injury, poisoning and procedural complications) | 1 (1)
Pain Below the Level of Implant (Injury, poisoning and procedural complications) | 2 (2)
Persistent Pain at The IPG Site (Injury, poisoning and procedural complications) | 1 (1)
Skin Erosion Around the Implant (Injury, poisoning and procedural complications) | 1 (1)
Skin Irritation at IPG Site (Injury, poisoning and procedural complications) | 1 (1)
Stimulation in Unwanted Places/Chest Wall Stimulation (Injury, poisoning and procedural complications) | 1 (1)
Weakness, Clumsiness, Numbness or Pain Below the Level of Implant (Injury, poisoning and procedural complications) | 1 (1)
Acute Appendicitis (Infections and infestations) | 1 (1)
Acute Renal Failure (Renal and urinary disorders) | 1 (1)
Aspiration Pneumonia (Infections and infestations) | 1 (1)
Bone Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis of Left Upper Extremity (Infections and infestations) | 1 (1)
Cerebral Infarction Due to Embolism of Unspecified Cerebral Artery (Nervous system disorders) | 1 (1)
Cholecystectomy (Hepatobiliary disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Death of Unknown Cause (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Heart Attack (Cardiac disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Staph Infection (Infections and infestations) | 1 (1)
Suicide Ideation (Psychiatric disorders) | 1 (1)
Syncope and Bleeding After Colonoscopy (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Subjects (N=269)
Broken Swift Lock Anchors (Injury, poisoning and procedural complications) | 1 (1)
Burning Pain at The IPG Site (Injury, poisoning and procedural complications) | 1 (1)
Cerebrospinal Fluid (CSF) Leakage (Injury, poisoning and procedural complications) | 2 (2)
Changes in Stimulation or Reduced Pain Relief Due to Lead Failure (Injury, poisoning and procedural complications) | 4 (4)
Changes in Stimulation or Reduced Pain Relief Due to Lead Migration (Injury, poisoning and procedural complications) | 4 (4)
Changes in Stimulation or Reduced Pain Relief Due to Loose Electrical Connections (Injury, poisoning and procedural complications) | 2 (2)
Chronic Pain Exacerbation Due to Battery Depletion (Injury, poisoning and procedural complications) | 1 (1)
Damage to Functionality/ Mechanical Integrity of IPG Resulting in Inability to Communicate with IPG (Injury, poisoning and procedural complications) | 2 (2)
Damage to IPG/Leads Causing System Fail Deliver Stimulation/Causing System Deliver Overstimulation (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Inadequate Stimulation (Injury, poisoning and procedural complications) | 1 (1)
Increased Pain (Injury, poisoning and procedural complications) | 1 (1)
Infection (Injury, poisoning and procedural complications) | 3 (3)
Insufficient Pain Relief (Injury, poisoning and procedural complications) | 1 (1)
Persistent Pain at The IPG Site (Injury, poisoning and procedural complications) | 3 (3)
Persistent Pain at The Lead Site (Injury, poisoning and procedural complications) | 1 (1)
Stimulation in Unwanted Places/Chest Wall Stimulation (Injury, poisoning and procedural complications) | 1 (1)
Undesirable Changes in Stimulation Which May Be Due to Cellular Changes in Tissue Around Electrodes (Injury, poisoning and procedural complications) | 1 (1)
Weakness, Clumsiness, Numbness or Pain Below the Level of Implant (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT03082261/Prot_SAP_001.pdf